CLINICAL TRIAL: NCT05171153
Title: Analysis of Bone Quality in Adult Patients With Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Quironsalud (Other)
Responsible Party: Principal Investigator, Maria Cortes, Endocrinology MD, Quironsalud
Other Study IDs: PIC108-21_HRJB
Record Dates: First submitted 2021-11-09; First posted 2021-12-28 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Inflammatory Bowel Diseases; Osteoporosis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Osteoporosis | interventions — Densitometry; Clinical Laboratory Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IBD group: Subjects over 21 years old, with inflammatory bowel disease (both ulcerative colitis and Crohn's disease), diagnosed by clinical, biochemical, endoscopic and anatomo-pathological criteria.
  Interventions: Other: Densitometry with Trabecular Bone Score; Other: Quantitative Ultrasound of Calcaneus; Other: Laboratory test
- Control group: Subjects over 21 years old, without IBD or known metabolic bone disease, recruited voluntarily in the Endocrinology and Nutrition, Digestive System and Rheumatology departments of the Ruber Juan Bravo Hospital, during routine health control visits
  Interventions: Other: Densitometry with Trabecular Bone Score; Other: Quantitative Ultrasound of Calcaneus; Other: Laboratory test

INTERVENTIONS:
Other: Densitometry with Trabecular Bone Score — Conventional bone densitometry at the level of the proximal femur and lumbar spine (L1-L4) (anteroposterior and lateral) measured with a General Electric Prodigy Advance Full enCORE version 11.x equipment. With the data from the lateral densitometry, and using the "VFA Dual Vertebral Assessment H8650DA/DM" software, a quantitative morphometric analysis of the thoracolumbar vertebrae (T4-L4) will be carried out. Additionally, microarchitectural parameters of the lumbar spine will be evaluated with TBS (iNsight v3.0) and bone quality in the proximal femur with the DEXA-3D 3D-SHAPER v2.10.1 software. Vertebral fracture will be excluded from the DXA and TBS analysis of the spine.
  Other Names: General Electric Prodigy Advance Full enCORE version 11.x
Other: Quantitative Ultrasound of Calcaneus — Quantitative bone ultrasound of calcaneus evaluated with a SONOST 3000, (OsteoSys Co, Korea).
  Other Names: Sonost 3000
Other: Laboratory test — Analysis of general biochemical parameters and serum phospho-calcium metabolism, including: total calcium, albumin, phosphorus, 25-OH-vitamin D, intact PTH (iPTH), creatinine, estimated glomerular filtration rate, carboxy-terminal telopeptide of type I collagen ß-CTx (Crosslaps) and N-terminal propeptide of type I procollagen (P1NP).

SUMMARY:
Inflammatory bowel disease (IBD) is considered a risk factor for the development of osteoporosis, which leads to an increased risk of fractures. There is no data on bone quality obtained with imaging techniques other than bone densitometry such as Trabecular Bone Score (TBS), 3D bone densitometry (DXA-3D) or quantitative bone ultrasound (QUS). The TBS study can provide information on bone microarchitecture in these patients, with TBS values expected to be lower than those of subjects without IBD, with a decrease of up to 50 points in this parameter.

Primary objective: to evaluate and compare TBS values in patients with IBD and in a control group of volunteers without IBD or known metabolic bone pathology, adjusted for age, sex and body mass index (BMI).

Secondary objectives: to evaluate and compare results in DEXA parameters, QUS, DEXA-3D, biochemical parameters and FRAX data between patients with IBD and controls. To evaluate the prevalence of vertebral fractures analyzed by VFA. As well as to evaluate the evolution in one year of all these parameters in patients with IBD.

Prospective observational study with a cohort of patients with IBD and another of volunteers without IBD or metabolic bone pathology, adjusted for age, sex and BMI. Baseline bone quality data will be analyzed by bone densitometry, TBS, DEXA-3D and QUS, fractures assessed by VFA and bone remodeling markers in both cohorts. Subsequently, a one-year analysis of the parameters of the IBD cohort will be performed.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is considered a risk factor for the development of osteoporosis, which leads to an increased risk of fractures. There is no data on bone quality obtained with imaging techniques other than bone densitometry such as Trabecular Bone Score (TBS), 3D bone densitometry (DXA-3D) or quantitative bone ultrasound (QUS).

HYPOTHESES OF THE STUDY Subjects with inflammatory bowel disease present an alteration in bone quality that can be assessed by TBS, with TBS values expected to be lower than those of subjects without IBD or known bone pathology, with a decrease of up to 50 points in this parameter.

Primary Objective : to evaluate and compare the values of the trabecular bone score (TBS), a surrogate marker of bone quality, in patients with inflammatory bowel disease (IBD) and in a control group of volunteers without IBD or known metabolic bone pathology, recruited in the consultations of the Endocrinology and Nutrition, Digestive System and Rheumatology departments of the Hospital Ruber Juan Bravo during routine health control visits, adjusted for age, sex and body mass index (BMI).

Secondary Objectives

1. To compare bone mineral density (BMD) values measured by dual energy X-ray absorptiometry (DXA) at the lumbar spine (anteroposterior and lateral) and proximal femur in patients with IBD with those of a control group of subjects adjusted for age, sex and BMI.
2. To compare the ultrasound velocity and attenuation parameters (BUA and SOS) obtained by quantitative ultrasound of the calcaneus (QUS) in patients with IBD with those of a control group of subjects adjusted for age, sex and BMI.
3. To analyse the prevalence and severity of vertebral fractures using the Vertebral Fracture Assessment (VFA) software of lateral DXA in patients with IBD compared to a control group adjusted for age, sex and BMI.
4. To correlate the TBS results with the ultrasound velocity and attenuation parameters (BUA and SOS) obtained with QUS.
5. To correlate TBS results with BMD parameters measured by DXA in the lumbar spine (anteroposterior and lateral) and in the proximal femur.
6. To compare biochemical markers of bone remodelling [carboxy-terminal telopeptide of type I collagen (ß-CTx Crosslaps) and N-terminal propeptide of type I protocolagen (P1NP)] in patients with IBD with a control group of subjects adjusted for age, sex and BMI.
7. To correlate baseline levels of biochemical markers of bone remodelling with the results of: a) BMD obtained with DXA in the lumbar spine (anteroposterior and lateral) and in the proximal femur, b) TBS values and c) parameters obtained with QUS.
8. To assess the absolute 10-year risk of major fractures and hip fractures using the FRAX tool, in subjects with IBD. To correlate the absolute risk of fractures with the TBS and QUS values.
9. To evaluate the effect of adjusting the FRAX tool by including TBS values for the calculation of the absolute risk of major and hip fractures.
10. To analyse the evolution of bone microarchitecture parameters measured by TBS, bone ultrasound parameters of ultrasound velocity and attenuation, BMD in the lumbar spine (anteroposterior and lateral) and in the proximal femur and biochemical markers of bone remodelling in patients with IBD after one year of follow-up.
11. To analyse the discriminative capacity for the diagnosis of vertebral fractures evaluated with VFA of the TBS and QUS values, compared with the BMD values obtained in lumbar DXA (anteroposterior and lateral) in patients with IBD.
12. To compare volumetric BMD parameters measured by 3D bone densitometry (DXA-3D) of the hip in patients with IBD with a control group of subjects adjusted for age, sex and BMI.
13. To correlate bone quality parameters measured by TBS and QUS with volumetric BMD measured by 3D DXA-3D in the hip.
14. To evaluate the effect of the different disease-modifying treatments (biologicals, corticoids, etc.) on TBS values, bone ultrasound parameters, BMD values by conventional DXA and DXA-3D in patients with IBD.

This study is organised into two sub-studies:

* Sub-study 1: observational, analytical, prospective, cross-sectional. Cohort-type study, with a cohort of patients with IBD and a cohort of volunteers without IBD or known metabolic bone pathology, recruited in the consultations of the Endocrinology and Nutrition, Digestive System and Rheumatology departments of the Ruber Juan Bravo Hospital during routine health control visits, adjusted for age, sex and body mass index (BMI). The baseline data on bone quality measured by: a) bone densitometry in the lumbar spine (anteroposterior and lateral), b) bone densitometry in the proximal femur, c) TBS, d) DEXA-3D, e) calcaneal ultrasound, e) fractures assessed by VFA and f) biochemical markers of bone remodelling in both cohorts will be analysed to respond to the primary objective, secondary objectives 2 to 9 and exploratory objectives 11 to 14.
* Sub-study 2: observational, analytical, prospective and longitudinal, with one-year follow-up of IBD patients only. Bone quality parameters measured by: a) bone densitometry in the lumbar spine (anteroposterior and lateral), b) bone densitometry in the proximal femur, c) TBS, d) DEXA-3D, e) calcaneal ultrasound, e) fractures assessed by VFA and f) biochemical markers of bone remodelling will be analysed to respond to secondary objective 10.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects over 21 years old, with inflammatory bowel disease (both ulcerative colitis and Crohn's disease), diagnosed by clinical, biochemical, endoscopic and anatomo-pathological criteria.
2. Subjects over 21 years old, without IBD or known metabolic bone pathology, recruited voluntarily in the Endocrinology and Nutrition, Digestive System and Rheumatology departments of the Ruber Juan Bravo Hospital, during routine health control visits (control group).
3. Subjects without language barriers, who expressed their willingness to cooperate in the follow-up and who gave their informed consent before entering the study.

Exclusion Criteria:

1. Other concomitant causes of metabolic bone disease: Paget's disease, severe chronic renal insufficiency (estimated glomerular filtration rate <30 ml/min/1.73m2), metastatic bone disease, multiple myeloma, Hypercalcemia > 11 mg/dl, period of immobilisation for more than 3 months in the previous year.
2. Pregnant women or women planning pregnancy during the recruitment and testing process.
3. Anatomical alteration of the right foot that may interfere with calcaneal ultrasound, including moderate-severe edema.
4. Patients on active treatment with antiresorptive drugs, osteoformers, or pharmacological doses (>50,000 units/month) of vitamin D3 (cholecalciferol).
5. Patients with a history of treatment with oral bisphosphonates, strontium ranelate or therapeutic doses of fluoride (>20 mg/day) for more than 3 months in the two years prior to the baseline visit, or for more than two years at any time in their life.
6. Patients who have received an intravenous bisphosphonate in the three years prior to the baseline visit.
7. Patients who have received denosumab within 6 months prior to the baseline visit.
8. Patients who have received calcitonin or a selective oestrogen receptor modulator in the 3 months prior to the baseline visit.
9. Participation at the time of recruitment in a clinical trial with medicinal products for the prevention or treatment of osteoporosis and/or IBD.

   Additional exclusion criteria for the control group:
10. Chronic diseases affecting bone metabolism, for example, active hyperthyroidism within the last 6 months, Cushing's syndrome, anorexia nervosa, early menopause, type 1 diabetes mellitus, poorly controlled type 2 diabetes mellitus of more than 5 years' duration or with microvascular complications, or primary hyperparathyroidism.
11. Active treatment with drugs that affect bone quality such as corticoids, oral anticoagulants, anti-estrogens (aromatase inhibitors and/or GnRH analogues), anti-androgens and anti-retroviral

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of the Endocrinology and Nutrition, Digestive System and Rheumatology departments of the Ruber Juan Bravo Hospital,
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Trabecular Bone Score | 1 year
  Trabecular bone score

SECONDARY OUTCOMES:
BMD | 1 year
  bone mineral density
BQI | 1 year
  bone quality index
VFA | 1 year
  Vertebral Fractures
ß-CTx | 1 year
  Bone marker β-CrossLaps
P1NP | 1 year
  Bone marker P1NP

OTHER OUTCOMES:
Volumetric BMD | 1 year
  volumetric BMD by 3D bone densitometry (DXA-3D)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cortes, Principal Investigator — Quironsalud
Locations (1):
- Hospital Ruber Juan Bravo, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No